CLINICAL TRIAL: NCT07014787
Title: EFFECT OF GRADES OF CHONDROMALACIA ON STATIC AND DYNAMIC BALANCE: CROSS-SECTIONAL STUDY
Brief Title: Assessing the Effect of Different Grades of Chondromalacia on Static and Dynamic Balance Using Biodex Balance System
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Selwan Khaled Mahmoud, Teaching Assistant, Cairo University
Other Study IDs: P.T.REC/012/005573
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Chondromalacia Patella
Keywords: Biodex balance system static and dynamic balance assessment of chondromalacia
MeSH Terms: conditions — Chondromalacia Patellae

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Control Group: Control group of 20 healthy patients Normal MRI Study
- grade I chondromalacia.: Experimental group of 20 patients with grade I chondromalacia Softening and swelling, intact surface Nearly normal (soft indentation and/or superficial fissures and cracks) Increased T2 signal intensity of morphologically normal cartilage
- grade II chondromalacia: Experimental group of 20 patients with grade II chondromalacia. Fragmentation and fissuring of articular cartilage affecting an area of less than 0.5 inches Abnormal (lesions extending to <50% of cartilage depth) A: Superficial partial-thickness cartilage defect <50% of total articular surface thickness B: Deep partial-thickness cartilage defect >50% of total articular surface thickness
- grade III chondromalacia: Experimental group of 20 patients with grade III chondromalacia Fragmentation and fissuring of articular cartilage affecting an area greater than 0.5 inches Severely abnormal (lesions extending >50% of cartilage depth, but not through subchondral bone) Full-thickness cartilage defect
- grade IV chondromalacia: Experimental group of 20 patients with grade IV chondromalacia Cartilage erosion to bone Lesions involving subchondral bone

SUMMARY:
The aim of this study is to investigate the effect of grades of chondromalacia on static and dynamic balance.

DETAILED DESCRIPTION:
Chondromalacia patellae is a very common disorder which is characterized by softening, swelling, fraying, fissuring, and erosion of hyaline cartilage overlying the patella. Patellar chondromalacia could be observed as a cause of patellofemoral pain, as well as in patients with osteoarthritis, in patients with knee trauma, or even in asymptomatic patients.

Balance, as an essential function in human daily life and activities, can be defined as central nervous system input. Postural control can be divided into static balance and dynamic balance; static balance controls the oscillation amplitude of the body, and dynamic balance uses the body's internal and external information to analyze factors that influence the stability of interference (Such as walking, pushing and pulling),and to maintain postural control. The perfect combination of static and dynamic balance is key to normal activities of the human daily life.

100 patients, 80 with different grades of chondromalacia (Grade I, II, III, IV) with 20 participants in each group and 20 healthy participants in the control group will be recruited for the study to assess the effect of different chondromalacia grades on static and dynamic balance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranged from 18 to 40 years old
2. groups include both males and females
3. Patients with Grade I, II, III and IV chondromalacia: Confirmation of diagnosis by MRI
4. BMI will be ranged from 19.0 to 29.0
5. Patients with Unilateral or bilateral chondromalacia.
6. Chronic cases for more than 3 months.
7. Positive sign of Knee pain according to patellar Grind Test

Exclusion Criteria:

1. patients have not undergone knee replacement.
2. patients have not done Intra-articular injection in the affected knee for the past 3 months.
3. Patients with rheumatoid arthritis or other inflammatory arthritis.
4. Patients with Vestibular disorders or neurological conditions.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 100 patients, 80 with different grades of chondromalacia (Grade I, II, III, IV) with 20 participants in each group and 20 healthy participants in the control group will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Measuring static and dynamic balance | up to four weeks
  Measuring static and dynamic balance using biodex balance system

CONTACTS AND LOCATIONS:
Overall Officials: Selwan Khaled Ayad, Teacher Assistant, Principal Investigator — Cairo University
Locations (1):
- Faculty of physical therapy Cairo University, Giza, Egypt